CLINICAL TRIAL: NCT00772187
Title: Intraoperative and Postoperative Analgesia for Laparoscopic Surgery.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dror Segal, M.D, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rambam2690CTIL
Record Dates: First submitted 2008-05-21; First posted 2008-10-15 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-07

CONDITIONS: Analgesia
Keywords: Laparoscopic surgery (general surgery).
MeSH Terms: conditions — Agnosia | interventions — Morphine; Anesthesia, General; Fentanyl

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): General anesthesia + I.V pca
  Interventions: Drug: general anesthesia (fentanyl)
- 2 (Experimental): General anesthesia + spinal analgesia + I.V pca
  Interventions: Drug: morphine; Drug: intrathecal analgesia (morphine)

INTERVENTIONS:
Drug: morphine — Single dose: 0.1-0.5 mg
  Arms: 2
Drug: intrathecal analgesia (morphine) — 0.1-0.5 mg of morphine
  Arms: 2
Drug: general anesthesia (fentanyl) — general anesthesia alone
  Arms: 1

SUMMARY:
Main Hypothesis: laparoscopic surgery is very painful to patient during and after surgery. We would like to compare different analgesic methods.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic (general) Surgery
* Age>18
* ASA<4
* Morning surgery

Exclusion Criteria:

* Patient refusal
* contra-indication for treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Good analgesic method with minimal side effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel, Israel